CLINICAL TRIAL: NCT01936025
Title: A Phase IIa, Dose-finding, Double-blind, Placebo-controlled, Double-dummy, Randomized, Eightfold Cross-over Study to Investigate the Glucose Lowering Effects of Dextromethorphan Alone or in Combination With Sitagliptin in Subjects With Type 2 Diabetes Mellitus (T2DM) After an Oral Glucose Tolerance Test
Brief Title: A Study to Investigate the Glucose Lowering Effects of Dextromethorphan Alone or in Combination With Sitagliptin in Subjects With Type 2 Diabetes Mellitus (T2DM) After an Oral Glucose Tolerance Test
Acronym: DXM2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00/0648-DXM2
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Dextromethorphan; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sitagliptin (Active Comparator): Placebo dextromethorphan + sitagliptin 100 mg
  Interventions: Drug: Sitagliptin
- Dextromethorphan 30 mg + sitagliptin (Experimental): Dextromethorphan 30 mg + sitagliptin 100 mg
  Interventions: Drug: Dextromethorphan; Drug: Sitagliptin
- Dextromethorphan 60 mg + sitagliptin (Experimental): Dextromethorphan 60 mg + sitagliptin 100 mg
  Interventions: Drug: Dextromethorphan; Drug: Sitagliptin
- Dextromethorphan 90 mg + sitagliptin (Experimental): Dextromethorphan 90 mg + sitagliptin 100 mg
  Interventions: Drug: Dextromethorphan; Drug: Sitagliptin
- Dextromethorphan 30 mg + placebo (Experimental): Dextromethorphan 30 mg + placebo (sitagliptin)
  Interventions: Drug: Dextromethorphan
- Dextromethorphan 60 mg + placebo (Experimental): Dextromethorphan 60 mg + placebo (sitagliptin)
  Interventions: Drug: Dextromethorphan
- Dextromethorphan 90 mg + placebo (Experimental): Dextromethorphan 90 mg + placebo (sitagliptin)
  Interventions: Drug: Dextromethorphan
- Placebo (Placebo Comparator): Placebo (dextromethorphan)+ placebo (sitagliptin)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan
  Arms: Dextromethorphan 30 mg + placebo; Dextromethorphan 30 mg + sitagliptin; Dextromethorphan 60 mg + placebo; Dextromethorphan 60 mg + sitagliptin; Dextromethorphan 90 mg + placebo; Dextromethorphan 90 mg + sitagliptin
Drug: Sitagliptin
  Arms: Dextromethorphan 30 mg + sitagliptin; Dextromethorphan 60 mg + sitagliptin; Dextromethorphan 90 mg + sitagliptin; Sitagliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study has a randomized, double-blind, placebo-controlled, double dummy and eight-way cross-over design. Males with T2DM on a stable metformin monotherapy will be screened for participation in the study. Eligible subjects will be randomized to receive DXM 30 mg, DXM 60 mg, DXM 90 mg alone or in combination with sitagliptin 100 mg, sitagliptin 100 mg alone, or placebo (for DXM and sitagliptin) on in total eight treatment days. An OGTT will be started 1 hour after study drug administration and blood glucose will be measured over the next 4 hours. There will be a 3 to 14-day washout period between doses.

DETAILED DESCRIPTION:
This study is performed to determine the optimal dose of DXM that, compared to placebo, decreases glucose excursions following an OGTT. Doses of 30 mg, 60 mg and 90 mg DXM were chosen. Since DXM 60 mg was effective in the previous study in increasing insulin secretion, this dose will be kept. A lower dose (30 mg) will be given to see whether effects on insulin secretion are present also at lower doses and then translate into a BG lowering action. A higher dose (90 mg) will be added to see whether this way an effect on glucose excursion reduction occurs following an OGTT, (like previously demonstrated with 270 mg DXM) that can be related to an increase of insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent obtained before any study-related activities
2. Male subjects with a diagnosis of type 2 diabetes mellitus according to ADA criteria at least 4 months prior to screening
3. Medical history without major pathology (with the exception of type 2 diabetes)
4. On a stable regimen of metformin monotherapy for at least 3 months
5. Aged between 45 and 70 years of age, both inclusive
6. Body mass index (BMI) between 25 and 35kg/m2, both inclusive

Exclusion Criteria:

1. Subjects with type 1 diabetes, MODY or secondary forms of diabetes such as due to pancreatitis
2. History of pancreatitis
3. Current or previous treatment with insulin therapy
4. Treatment with any hypoglycemic medication other than metformin within the three months prior to screening
5. Mean QTc> 450 msec

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
lowest dose of DXM | up to 4 hours after study drug administration
  To find the lowest dose of DXM that, compared to placebo, exerts BG lowering effects related to an OGTT

SECONDARY OUTCOMES:
additive BG lowering effects | up to 4 hours after study drug administration
  To demonstrate whether the administration of DXM on top of sitagliptin exerts additive BG lowering effects related to an OGTT as compared to sitagliptin alone and DXM alone

CONTACTS AND LOCATIONS:
Overall Officials: Alin Stirban, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Marquard J, Stirban A, Schliess F, Sievers F, Welters A, Otter S, Fischer A, Wnendt S, Meissner T, Heise T, Lammert E. Effects of dextromethorphan as add-on to sitagliptin on blood glucose and serum insulin concentrations in individuals with type 2 diabetes mellitus: a randomized, placebo-controlled, double-blinded, multiple crossover, single-dose clinical trial. Diabetes Obes Metab. 2016 Jan;18(1):100-3. doi: 10.1111/dom.12576. Epub 2015 Oct 26. PMID 26362564